CLINICAL TRIAL: NCT02466828
Title: Quantitative Blood Oxygenation Level Dependent (qBOLD) MR Imaging of Glioblastoma Multiforme for Assessment of Tumor Hypoxia.
Brief Title: qBOLD MRI of Glioblastoma Multiforme for Assessment of Tumor Hypoxia.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 127-2014
Record Dates: First submitted 2014-11-21; First posted 2015-06-09 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Glioblastoma; Hypoxia
MeSH Terms: conditions — Glioblastoma; Hypoxia | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single patient group receiving Feraheme® (Experimental): Newly diagnosed GBM patients with no prior treatment will receive Feraheme® as MRI contrast agent
  Interventions: Drug: Feraheme®

INTERVENTIONS:
Drug: Feraheme® — Drug will be diluted in 50 cc normal saline and infused over 15-60 minutes depending on patient condition.
  Other Names: ferumoxytol

SUMMARY:
Glioblastoma multiforme (GBM) is the most common primary malignant brain neoplasm in adults. Despite recent diagnostic and therapeutic advances, including aggressive surgical resection and chemoradiation, the prognosis of GBM has improved only slightly over the past two decades, with median survival of approximately 15 months. Tumor hypoxia is a feature of GBM that contributes to poor outcome through multiple mechanisms such as 1) overexpression of enzymes that play roles in temozolomide resistance, the main chemotherapeutic agent in GBM and 2) increase expression of cancer stem cells which are more resistant to radiation. Hypoxic tumour regions are associated with higher rates of progression and recurrence.

In this study the investigators will use an advanced MRI technique called qBOLD to non-invasively measure oxygenation in GBM and obtain targeted biopsies. The investigators take advantage of physical characteristics of Ferumoxytol (Feraheme®) which is an iron supplement, and utilize two recent technical advances not previously used in human tumours to quantitatively measure oxygenation in GBM.

Prior knowledge of hypoxia can assist in prognostication and individualization of treatment planning with special focus on hypoxic regions by targeted radiation dose or regimen modulation; consideration of more intensive chemotherapy regimens; more aggressive and targeted surgical resection and closer short-term clinical and imaging follow-ups.

DETAILED DESCRIPTION:
We propose a study to demonstrate quantitative oxygen saturation estimation in GBM is feasible with qBOLD and it correlates with established histopathological markers of hypoxia and angiogenesis, and targeted intraoperative oxygen measurement.

All patients will undergo surgery as part of their standard treatment. By coregistering the hypoxia map on presurgical MRI we will be able to do the following:

1. Obtain targeted biopsies of the hypoxic areas and none hypoxic areas and correlate them with gold standard marker of tissue hypoxia by immunohistochemistry for hypoxia induced factor-1α (HIF-1α).
2. Draw Volumes of interests (VOI) over areas >0.5-cm3 (amenable to accurate intra-operative O2 measurement) with the lowest and highest oxygen saturation (SO2) values. VOIs will be then imported into the neuronavigation system (Stryker) for targeted placement of clinically approved Licox® oxygen-sensing probe (Integra NeuroSciences).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 year old) patients with newly diagnosed GBM presenting to our centre for surgical management and post-operative chemoradiation
2. Creatinine clearance > 60 ml/minute
3. Able to tolerate an MR scan
4. Capable of providing informed consent.

Exclusion Criteria:

1. Prior brain surgery or radiation
2. History of liver disease requiring liver MRI (due to accumulation of ferumoxytol in Kupffer cells which can affect liver MRI for up to 3 months)
3. On more than two antihypertensive medications
4. History of allergy or adverse reaction to iron supplements
5. Prior treatment with ferumoxytol
6. Large (>50%) hemorrhagic component in the solid enhancing part of the tumor
7. Need for emergency craniotomy.
8. Pregnant patients
9. Breast feeding
10. Serum ferritin of >800 ng/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation in GBM with qBOLD MRI and its correlation with histological markers of tissue hypoxia and angiogenesis | Within 8 hours after the MRI exam is complete
  Pre-operative qBOLD imaging and O2 saturation mapping will be performed in 27 newly diagnosed GBM patients and targeted biopsies will be obtained from the hypoxic and non-hypoxic regions of the tumor.

SECONDARY OUTCOMES:
Oxygen saturation in GBM with qBOLD MRI and its correlation with targeted intraoperative oxygen measurement | Within 8 hours after the MRI exam is complete
  Volumes of interest from the hypoxic and non-hypoxic regions of the tumor will be imported into the neuronavigation system (Stryker) for targeted placement of Licox® oxygen-sensing probe (Integra NeuroSciences).

CONTACTS AND LOCATIONS:
Overall Officials: Pejman Jabehdar Maralani, MD FRCPC, Principal Investigator — Sunnybrook Health Sciences Center
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario